CLINICAL TRIAL: NCT02135705
Title: LOWER: Lomitapide Observational Worldwide Evaluation Registry
Acronym: LOWER
Status: Recruiting | Type: Observational
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: AEGR-733-025
Record Dates: First submitted 2014-04-10; First posted 2014-05-12 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lomitapide: Lomitapide as prescribed by Physician.
  Interventions: Drug: Lomitapide

INTERVENTIONS:
Drug: Lomitapide — As prescribed by Physician.
  Other Names: Juxtapid; Lojuxta

SUMMARY:
This global product exposure registry is a multicentre, long-term, prospective, observational cohort study (exposure registry), designed to evaluate the long term safety and effectiveness of lomitapide.

DETAILED DESCRIPTION:
To evaluate the occurrence of adverse events of special interest, long term effectiveness of lomitapide, and to evaluate whether prescribers of lomitapide are following screening and monitoring recommendations as specified in product labeling.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages, including minors, who have initiated commercial treatment with lomitapide prior to or at time of registry enrolment.
* Patients who have the ability to understand the requirements of the study and provide written informed consent to comply with the study data collection procedures or paediatric patients with the consent of a parent or legal guardian.

Patients ≥7 years of age (or above the age determined by the IRB/EC and in accordance with the local regulations and requirements) must also provide written informed assent forms.

Exclusion Criteria:

* Patients who are receiving lomitapide in clinical trials or through compassionate use, where patients are followed under a separate protocol.
* Patients receiving an investigational agent, defined as any drug or biologic agent other than lomitapide that has not received market authorization in the country of participation, at time of lomitapide initiation and continuing to receive an investigational agent at time of registry enrolment. These patients may be enrolled if receiving lomitapide when the investigational agent is discontinued..

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with lomitapide who agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-03-18 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Hepatic Abnormalities | patients will be followed for 10 years
  to evaluate the occurrence of hepatic abnormalities

SECONDARY OUTCOMES:
Gastrointestinal (GI) Events | patients will be followed for 10 years
  to evaluate the occurrence of GI events
Tumors | patients will be followed for 10 years
  to evaluate any occurrence of tumors (small bowel, hepatic, colorectal or pancreatic)
Events associated with coagulopathy | patients will be followed for 10 years
  to evaluate the occurrence of events associated with coagulopathy (abnormal bleeding, cerebral haemorrhage or GI bleeding)
Major Adverse Cardiovascular Events (MACE) events | patients will be followed for 10 years
  to evaluate the occurrence of MACE events
Death, including cause of death | patients will be followed for 10 years
  to evaluate the occurrence and cause of death
Pregnancy | patients will be followed for 10 years
  to evaluate the occurrence and outcomes of pregnancy in females of reproductive potential treated with lomitapide. Patients who become pregnant will be offered enrolment into a separate Pregnancy Exposure Registry (PER).
Serum lipid levels | patients will be followed for 10 years
  to evaluate the long-term effectiveness of lomitapide in maintaining control of serum lipid levels in a clinical practice setting.
Prescriber behavior | patients will be followed for 10 years
  to evaluate whether prescribers of lomitapide enrolled at registry sites are following the screening and monitoring recommendations as specified in the PI and the prescriber educational materials aimed at risk minimization.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Boylan, Study Director — Amryt Pharmaceuticals
Locations (75):
- United States (50):
  - Brookwood Baptist Medical Center, Birmingham, Alabama
  - Springhill Physician Practices, Mobile, Alabama
  - Northern Arizona Healthcare, Cottonwood, Arizona
  - One Medical, Gilbert, Arizona
  - Scottsdale Family Health, Phoenix, Arizona
  - Pima Heart, Tucson, Arizona
  - Arkansas Heart Center, Fort Smith, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Health, Aurora, Colorado
  - Alfieri Cardiology, Newark, Delaware
  - Preventative Cardiology, Inc., Boca Raton, Florida
  - Florida Lipid Institute, Winter Park, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Atlanta Heart Specialists, Cumming, Georgia
  - Northside Hospital, Inc., Cumming, Georgia
  - Comprehensive Cardiovascular Care, Gurnee, Illinois
  - Community Health Network, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - Henry County Medical Center, New Castle, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Get Well Immediate Care, Towson, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Complete Family Care Cholesterol Treatment Center, Sterling Heights, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - HealthEast Care System, Saint Paul, Minnesota
  - Stern Cardiovascular Foundation, Southaven, Mississippi
  - Methodist Physicians Clinic, Omaha, Nebraska
  - Hackensack Meridian Health, Edison, New Jersey
  - Avinash C. Gupta, MD, PC, Lakewood, New Jersey
  - 201 Route 17 North, Rutherford, New Jersey
  - Valley Medical Group, Wyckoff, New Jersey
  - Murray Hill Medical Group, New York, New York
  - NY Heart Center, Syracuse, New York
  - Pediatric Cardiology Associates, Syracuse, New York
  - Cardiology Specialists of the Carolinas PA, Charlotte, North Carolina
  - Cardiology Specialists Of Carolina, Charlotte, North Carolina
  - The Heart Care Group, PC, Allentown, Pennsylvania
  - St. Luke's University Health Network - Pennsylvania, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital And Health Network, East Stroudsburg, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Health System, Philadelphia, Pennsylvania
  - Palmetto Health, Columbia, South Carolina
  - 317 Saint Francis Dr., Greenville, South Carolina
  - Cardiovascular Specialists of Texas, Austin, Texas
  - Baylor Scott & White Health, Dallas, Texas
  - The University of Vermont Health Network, Burlington, Vermont
  - West Virginia University Medicine, Morgantown, West Virginia
  - Ascension, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aspirus Research Institute, Wausau, Wisconsin
- Clinica de Salud de Chaco, Reconquista, Chaco CPA, Argentina
- Canada (4):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Robarts Research Institute, London, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - McGill University, Montreal, Quebec
- France (3):
  - Centre Hospitalier Régional Universitaire de Lille, Lille, Cedex
  - Centre Hospitalier Universitaire Lyon, Bron, Lyon
  - Centre Hospitalier Universitaire Strasbourg, Strasbourg
- Greece (2):
  - University General Hospital of Ioannina, Ioannina
  - Metropolitan Hospital, Piraeus
- Italy (12):
  - Policlinico S. Orsola-Malpighi, Bologna, BO
  - Azienda Ospedaliera G. Brotzu, Cagliari, CA
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, PA
  - Azienda Ospedaliera Universita di Padova, Padua, PD
  - Università degli Studi di Roma La Sapienza, Roma, RM
  - Università degli Studi di Roma La Sapienza, Roma, Rome
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, TO
  - Azienda Ospedaliero Universi consorziale policlinico di Bari, Bari
  - Azienda Ospedaliera Specialistica Dei Colli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - CNR Regione Toscana - Fondazione Toscana Gabriele Monasterio, Pisa
- Netherlands (2):
  - Radboud Universiteit Medisch Centrum, Nijmegen, Gelderland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
- Imperial College Healthcare - NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Larrey D, D'Erasmo L, O'Brien S, Arca M; Italian Working Group on Lomitapide. Long-term hepatic safety of lomitapide in homozygous familial hypercholesterolaemia. Liver Int. 2023 Feb;43(2):413-423. doi: 10.1111/liv.15497. Epub 2022 Dec 30. PMID 36520008
- [Derived] Giammanco A, Cefalu AB, Noto D, Averna MR. Therapeutic Options for Homozygous Familial Hypercholesterolemia: The Role of Lomitapide. Curr Med Chem. 2020;27(23):3773-3783. doi: 10.2174/0929867326666190121120735. PMID 30663562